CLINICAL TRIAL: NCT02165241
Title: Characterization of the Immunological Profile in Relation to Cardiac Geometry Variations in Hypertensive Patients
Brief Title: Immunological Profile in Relation to Cardiac Geometry in Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Giuseppe Lembo, Professor, MD, PhD, Neuromed IRCCS
Other Study IDs: LMB01
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Immune System Profile During Hypertensive Cardiac Remodeling
Keywords: Hypertension; Cardiac remodeling; Immune system
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
It is commonly known that heart failure (HF) is the main cause of mortality and morbidity which affects about 15 million people in the world and is the primary chronic cause of death. In spite of the development of pharmacological therapies which have led to a good control of the pathology, almost 50% of patients with advanced HF does not survive after the first year. Heart failure consists of a deterioration of the cardiac pump, whose performance become insufficient to satisfy the organism needs. HF can be the consequence of various pathologies, such as ischemia, chronic hypertension, valvulopathies, pericarditis, etc. In conditions of chronic overload, as the one induced by the cited pathologies, the cardiomyocytes reply with hypertrophy and/or death due to necrosis or apoptosis. At the same time, there is a collagen alteration which causes the substitution of the myocardial damaged portion with fibrotic material, increasing in this way cardiac rigidity and reducing contractility. Finally, the onset of inflammation, the activation of the immune system and of the inflammatory mediators affect heart functionality. These phenomena are regulated by a complex interaction between the cellular and molecular mechanisms, which moreover guarantee the homeostasis maintenance in physiological conditions. Nevertheless, their imbalance activates a complex series of events which have recently started to be recognized and studied. In effect, a recent work has underlined the importance of the splenic monocytes in the cardiac response to acute heart ischemia, changing our vision concerning the role of the immune system in heart diseases.Historically, the term "cardiac remodeling" had been introduced to describe the anatomical change of the heart which occurs after myocardial infarction. At a later stage, it has been acknowledged that also other pathological conditions, such as chronic hypertension, can be a cause of the myocardial remodeling. Physiologically, the immune system cells have always been considered for their role of protection from infections. Recently, instead, evidence have been showing that immune system cells might have far more complex functions in the heart. The myocardial remodeling comes from modifications that may be adaptive to the initial insult, but then this structural adjustment may become the activation of structural/metabolic circles which can potentially culminate in the transition to HF.

This observational study will evaluate the immunological profile in relation to cardiac geometry variations in hypertensive patients. Aim of this project is to characterize the profile of immune system activation during the process of cardiac remodeling which is typical of the cardiomyopathy of overload. The main goal will be reached through the characterization of the circulating profile of immune system cells, in order to find a correlation with the clinical phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients between 30 and 65 years of age
* Subjects with a new diagnosis of hypertension not in treatment OR Subjects on antihypertensive treatment in need of further diagnostic analysis to evaluate the possibility of secondary hypertension. In this case treatment suspension will be necessary in order to obtain the ideal conditions for a diagnostic evaluation, in accordance with the guidelines for the management of arterial hypertension.
* Absence of cardiac remodeling at the echocardiographic examination
* Written informed consent prior to enrollment in the study

Exclusion Criteria:

* precedent acute myocardial infarction (AMI)
* unstabile angina
* congestive heart failure
* hemodynamically significant valvulopathies
* peripheric vasculopathies
* atrioventricular conduction diseases
* history of atrial fibrillation or other severe arrythmias
* malignant hypertension (200/140 mmHg)
* renal pathologies (creatinine > 1.4 mg/dL)
* severe respiratory diseases (COPD and allergic asthma)
* autoimmune disorders
* inflammatory diseases or patients with anti-inflammatory therapies
* diabetes mellitus
* previous and/or concomitant tumors
* anemia (haemoglobin <10g%)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the outpatient cardiac centre of the IRCCS Mediterranean Neurological Institute Neuromed, according to specific inclusion criteria. Approximately 100 subjects aged between 30 and 65 years will be included in the study. At the present 30 subjects have been enrolled.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Cardiac Remodeling | 24 months
  Changes in left ventricular (LV) posterior wall thickness; intraventricular septum thickness (IVS); LV diameter (LVD) and Relative Wall Thickness (RWT)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, (IS), Italy